CLINICAL TRIAL: NCT01160198
Title: A Multicentre, Randomized, Laboratory-blinded, Parallel-group Study to Demonstrate the Efficacy and Tolerability of Ferrous Bisglycinate Chelate in Iron Deficiency Anaemia and to Compare These With Those of Ferrous Ascorbate.
Brief Title: A Study to Demonstrate the Efficacy and Tolerability of Ferrous Bisglycinate Chelate in Iron Deficiency Anaemia and to Compare These With Those of Ferrous Ascorbate.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 114204
Record Dates: First submitted 2010-07-01; First posted 2010-07-12 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2017-09

CONDITIONS: Haematopoiesis
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ferrous bisglycinate chelate 1 OD (Experimental): ferrous bisglycinate chelate 1 tablet daily
  Interventions: Dietary Supplement: ferrous bisglycinate chelate 1 OD
- ferrous ascorbate (Active Comparator): ferrous ascorbate, 1 tablet daily
  Interventions: Drug: ferrous ascorbate
- ferrous bisglycinate chelate 2 OD (Experimental): ferrous bisglycinate chelate 2 tablets daily
  Interventions: Dietary Supplement: ferrous bisglycinate chelate 2 OD

INTERVENTIONS:
Drug: ferrous ascorbate — 100 mg elemental iron
  Arms: ferrous ascorbate
Dietary Supplement: ferrous bisglycinate chelate 1 OD — 60 mg elemental iron
  Arms: ferrous bisglycinate chelate 1 OD
Dietary Supplement: ferrous bisglycinate chelate 2 OD — 120 mg elemental iron
  Arms: ferrous bisglycinate chelate 2 OD

SUMMARY:
Iron deficiency anaemia (Haemoglobin, Hb < 12gm/dl) is one of India's major public health problems particularly in women. Effective control of iron deficiency anaemia decreases the incidence of fatigue, bodyache, headache, lack of concentration and menstrual complications. Iron bisglycine chelate has been used successfully to treat iron deficiency anaemia and is also a well tolerated therapy. Use of ferrous bisglycinate chelate one tablet daily as a nutritional supplement is well established in India. For treatment of iron deficiency anaemia, some women may need 1 tablet/day, while some may need 2 tablets/day. In India, ferrous ascorbate, 1 tablet daily is a widely accepted form of treatment for iron deficiency anaemia. The primary purpose of this study is to demonstrate the efficacy and tolerability profile of ferrous bisglycinate chelate to support the registration of this product as a 'drug' in India. Comparative data between ferrous bisglycinate chelate and ferrous ascorbate will also augment our existing knowledge, which will further support appropriate use of ferrous bisglycinate chelate for the treatment of iron deficiency anaemia. Study design and patient population: This will be a multicentre, randomized, laboratory-blinded, parallel- group study. It is projected that the study will randomize 270 women (90 subjects in each treatment arm) with iron deficiency anaemia (Hb 6-9 gm/dl + serum Ferritin <15 μg/l) to either ferrous bisglycinate chelate 1 or 2 tablets/day, or ferrous ascorbate 1 tablet/day for 8 weeks. At fortnightly visits, blood will be collected for Hb (to evaluate efficacy), adverse events will be documented (to evaluate tolerability), the investigational drugs will be dispensed and reasons for non compliance will be recorded. Study endpoints: The primary endpoint is defined as the rise of Hb from baseline after 8 weeks of treatment in each ferrous bisglycinate chelate group (1 tablet/day and 2 tablets/day). The secondary endpoints include the difference in the average change in Hb, difference in the rate of rise of Hb, difference in the proportion of patients who achieve a target Hb ≥12gm/dl and difference in the % incidence of gastrointestinal side effects during 8 week therapy with 2 dosing regimens of ferrous bisglycinate chelate (1 tablet/day and 2 tablets/day) and ferrous ascorbate 1 tablet/day.

DETAILED DESCRIPTION:
Rationale Iron deficiency is the most common form of malnutrition globally. In India, nearly 70% of women are estimated to be iron deficient. Iron deficiency anemia (IDA, Hb <12gm/dl) is a very late manifestation of iron deficiency. IDA is a consequence of decreased iron intake, increased iron loss from the body or increased iron requirements Blood loss during menstruation can predispose women to have poor iron stores and the presence of excess menstrual bleeding can contribute to the development of IDA in women. Patients with IDA usually present with fatigue, headache, bodyache, paraesthesia and lack of concentration. IDA can cause menorrhagia, which in turn can aggravate IDA. With severe anemia, there may be amenorrhoea as well.

Iron deficiency anaemia is often treated with iron tablets such as ferrous sulphate, ferrous fumarate and ferrous gluconate. It usually takes about 6-10 weeks for Hb to return to normal after initiation of oral iron therapy. Although efficacious from a haematological point of view, most of these therapies are associated with limiting gastrointestinal side effects (e.g. nausea, vomiting, constipation, diarrhoea and abdominal pain), which eventually reduce patient compliance.

Among the recent alternatives, iron bisglycine chelate has been used successfully to treat iron deficiency anaemia and is also a well tolerated therapy.

Use of ferrous bisglycinate chelate (each tablet contains 60mg of elemental iron as ferrous bisglycinate chelate, 1 mg folic acid, 5 mcg cyanocobalamin and 15 mg zinc bis-glycinate), 1 tablet daily is well established as a nutritional supplement in India. However, for treatment of iron deficiency anaemia, some women may need 1 tablet/day, while some may need 2 tablets /day.

In India, ferrous ascorbate tablets (each tablet contains 100 mg elemental iron as ferrous ascorbate, with 1 mg folic acid) in the recommended dose of 1 tablet daily are a widely accepted form of treatment for iron deficiency anaemia.

The primary purpose of this study is to demonstrate the efficacy and tolerability profile of ferrous bisglycinate chelate to support the registration of this product as a 'drug' in India. Comparative data between ferrous bisglycinate chelate and ferrous ascorbate will also augment our existing knowledge, which will further support the use of ferrous bisglycinate chelate for the treatment of iron deficiency anaemia.

Objective(s)

Primary:

To estimate the mean rise in haemoglobin level in patients with iron deficiency anaemia after 8 weeks of treatment (vs. baseline) with ferrous bisglycinate chelate (1 tablet and 2 tablets daily).

Secondary:

1. To compare the mean rise in haemoglobin in patients with iron deficiency anaemia after 8 weeks treatment with ferrous bisglycinate chelate, 1 tablet and 2 tablets daily vs. ferrous ascorbate 1 tablet daily.
2. To compare the average rate of rise of haemoglobin during 8 weeks of treatment with ferrous bisglycinate chelate 1 tablet daily, ferrous bisglycinate chelate 2 tablets daily and ferrous ascorbate 1 tablet daily.
3. To compare the proportion of patients who achieve a target Hb ≥ 12gm/dl after 8 weeks of treatment with ferrous bisglycinate chelate 1 tablet daily, ferrous bisglycinate chelate 2 tablets daily and ferrous ascorbate 1 tablet daily.
4. To compare the % incidence of gastrointestinal side effects during 8 weeks treatment with ferrous bisglycinate chelate 1 tablet daily, ferrous bisglycinate chelate 2 tablets daily and ferrous ascorbate 1 tablet daily.

Study Design This will be a multicentre, randomized, laboratory-blinded, parallel-group study. It is projected that the study will randomize 270 women (90 subjects in each treatment arm) with iron deficiency anaemia (Hb 6-9 gm/dl + serum Ferritin <15 μg/l) to either ferrous bisglycinate chelate 1 tablet/day, ferrous bisglycinate chelate 2 tablets/day or ferrous ascorbate 1 tablet/day for 8 weeks. At fortnightly visits, blood will be collected for Hb (to evaluate efficacy), adverse events will be documented (to evaluate tolerability), the investigational drugs will be dispensed and reasons for non compliance will be recorded.

The total study duration consists of an 8-week treatment period and will involve 6 clinic visits.

Study Endpoints/Assessments Primary Endpoint(s) Rise of haemoglobin from baseline to 8 weeks in each ferrous bisglycinate chelate group (1 tablet daily and 2 tablets daily).

Secondary Endpoint(s)

1. The difference in the average change in Hb from baseline to 8 weeks with ferrous bisglycinate chelate 1 and 2 tablets daily, and ferrous ascorbate 1 tablet daily.
2. The difference in the average rate of rise of Hb during 8 weeks of treatment with ferrous bisglycinate chelate 1 tablet daily, ferrous bisglycinate chelate 2 tablets daily, and ferrous ascorbate 1 tablet daily.
3. The difference in proportion of patients who achieve a target Hb ≥12gm/dl after 8 weeks of treatment with ferrous bisglycinate chelate 1 tablet daily, ferrous bisglycinate chelate 2 tablets daily, and ferrous ascorbate 1 tablet daily.
4. The difference in % incidence of gastrointestinal side effects during 8 weeks treatment with ferrous bisglycinate chelate 1 tablet daily, ferrous bisglycinate chelate 2 tablets daily and ferrous ascorbate 1 tablet daily.

ELIGIBILITY:
Inclusion Criteria

Subjects eligible for enrolment to the study must meet all of the following criteria:

1. Signed and dated written informed consent is obtained prior to participation.
2. Female outpatients between 18 to 55 years of age and using effective method of contraception if sexually active.
3. Non use of any iron supplement for 3 months prior to enrolment to the study.
4. Presence of iron deficiency anaemia: low haemoglobin (Hb 6-9 gm/dl) + low serum ferritin (<15 μg/l).
5. No occult blood in stool.
6. Able to comply with the requirements of the protocol.
7. Subjects should have a valid telephone contact.

Exclusion Criteria

Subjects meeting any of the following criteria must not be enrolled to the study:

1. Pregnancy (confirmed by urine dipstick method)
2. Desire to conceive within the next 3 months including patients who are receiving treatment to facilitate conception.
3. Lactating women.
4. Medical history of current hematological disorders other than iron deficiency anaemia (e.g. aplastic anaemia, megaloblastic anaemia, sideroblastic anaemia, pernicious anaemia, thalassemia, sickle cell anaemia, etc.).
5. Medical history of thyroid dysfunction.
6. Medical history of chronic renal disease.
7. Medical history of malabsorption syndrome, haemochromatosis and haemosiderosis, hypochlorhydria, achlorhydria, gastrectomy, gastrojejunostomy.
8. Inability to withhold prohibited medication.
9. Obvious internal or external bleeding as documented by medical history and/or examination if considered clinically significant in the opinion of the investigator.
10. Clinically significant abnormality in laboratory reports and/or ECG.
11. Medical history of hepatitis B, hepatitis C and/or exposure to HIV.
12. Serious, uncontrolled disease (other than thyroid dysfunction and chronic renal disease) including serious psychological disorders likely to interfere with the study and/or likely to cause death within the study period.
13. Participation in another clinical trial in the last 8 weeks before entry to Visit 0.
14. Evidence of alcohol or drug abuse, that may, in the opinion of the investigator interfere with study compliance or prevent understanding of the objectives, investigational procedures or possible consequences of the study.
15. Known or suspected hypersensitivity to iron or any of the components of ferrous bisglycinate chelate or ferrous ascorbate tablets.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2010-10-13 (Actual); Primary Completion 2011-02-18 (Actual); Study Completion 2011-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- India (6):
  - GSK Investigational Site, Bhojipura, Bareilly
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Surat
  - GSK Investigational Site, Thane,Mumbai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 centers in India from 12-October-2010 to 17-February-2011. OROFER XT™ (ferrous ascorbate, 100 milligram [mg]) is a registered product of Emcure Pharmaceuticals Ltd., Pune and Ferronine™ (ferrous bisglycinate chelate, 60 mg) is registered product of GlaxoSmithKline.
Pre-assignment Details: A total of 317 participants with iron deficiency anaemia were screened for this study; of these, 270 participants were randomized. Intent-to-Treat (ITT) population: all randomized participants who received at least one dose of study medication (n=270). Before randomization, all participants were dewormed with a single tablet of 400 mg albendazole.
Groups:
- Ferrous Bisglycinate Chelate 60 mg 1 Once-daily: Participants received ferrous bisglycinate chelate, 1 tablet of 60 mg, once-daily after dinner, via oral route for 8 weeks.
- Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily: Participants received ferrous bisglycinate chelate, 1 tablet each of 60 mg, twice-daily after breakfast and dinner, via oral route for 8 weeks.
- Ferrous Ascorbate 100 mg 1 Once-daily: Participants received ferrous ascorbate, 1 tablet of 100 mg once-daily after dinner, via oral route for 8 weeks.
Period: Overall Study
Arm/Group | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily | Ferrous Ascorbate 100 mg 1 Once-daily
Started | 89 | 91 | 90
Completed | 87 | 88 | 89
Not Completed | 2 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Participant lost drug; withdrew consent | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily | Ferrous Ascorbate 100 mg 1 Once-daily | Total
Number analyzed (Participants) | 89 | 91 | 90 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 89 | 91 | 90 | 270
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 91 | 90 | 270
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  India | 89 | 91 | 90 | 270

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hb) After 8 Weeks of Treatment in Each Ferrous Bisglycinate Chelate Group (1 Tablet Daily and 2 Tablets Daily)
Description: At fortnightly visits, blood was collected for Hb. Baseline (Visit 0) was not more than 5 days from Week 1 or randomization. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline and Week 8
Population: Per protocol (PP) population.
Measure: Mean (95% Confidence Interval); unit: Gram per deciliter (gm/dL)
Arm/Group | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily
Number analyzed (Participants) | 82 | 83
Gram per deciliter (gm/dL) | 2.6 [2.12 to 3.03] | 2.8 [2.36 to 3.31]
Statistical Analysis 1: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily; Baseline Hb vs. Hb at Week 8 for Ferrous bisglycinate chelate 60 mg 1 once-daily; Test type: Superiority or Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily; Baseline Hb vs. Hb at Week 8 for Ferrous bisglycinate chelate 60 mg 1 twice-daily; Test type: Superiority or Other; p < 0.0001, Paired t-test

2. Secondary Outcome: Mean Change in Hb From Baseline to 8 Weeks
Description: as for outcome 1
Time Frame: Baseline to Week 8
Population: PP population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (95% Confidence Interval); unit: gm/dL
Arm/Group | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily | Ferrous Ascorbate 100 mg 1 Once-daily
Number analyzed (Participants) | 82 | 83 | 87
gm/dL | 2.6 [2.12 to 3.03] | 2.8 [2.36 to 3.31] | 2.6 [2.19 to 3.09]

3. Secondary Outcome: Percentage of Participants Who Achieved a Target Hb More Than or Equal to 12 gm/dL After 8 Weeks of Treatment
Description: At fortnightly visits, blood was collected for Hb. Number of participants who achieved a target Hb of more than or equal to 12 gm/dL is presented.
Time Frame: Up to Week 8
Population: PP population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily | Ferrous Ascorbate 100 mg 1 Once-daily
Number analyzed (Participants) | 82 | 83 | 87
Percentage of participants | 34.2 | 36.1 | 33.3
Statistical Analysis 1: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous bisglycinate chelate 60 mg 1 twice-daily; Test type: Superiority or Other; p = 0.788, Chi-squared
Statistical Analysis 2: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous ascorbate 100mg 1 once-daily; Test type: Superiority or Other; p = 0.911, Chi-squared
Statistical Analysis 3: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 twice-daily vs. Ferrous ascorbate 100mg 1 once-daily; Test type: Superiority or Other; p = 0.700, Chi-squared

4. Secondary Outcome: Mean Change in Hb During 8 Weeks Therapy
Description: At fortnightly visits, blood was collected for Hb. Mean change in Hb at Week 2, Week 4, Week 6 and Week 8 are presented.
Time Frame: Up to Week 8
Population: PP population. Only those participants available at the specified time points were analyzed.
Measure: Mean (95% Confidence Interval); unit: gm/dL
Arm/Group | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily | Ferrous Ascorbate 100 mg 1 Once-daily
Number analyzed (Participants) | 82 | 83 | 87
gm/dL
  Week 2: number analyzed (Participants) | 81 | 83 | 87
  Week 2 | 0.6 [0.46 to 0.69] | 0.6 [0.50 to 0.78] | 0.7 [0.57 to 0.84]
  Week 4 | 1.2 [0.98 to 1.45] | 1.3 [1.07 to 1.61] | 1.4 [1.10 to 1.61]
  Week 6 | 1.8 [1.46 to 2.15] | 1.9 [1.58 to 2.32] | 1.9 [1.56 to 2.23]
  Week 8 | 2.6 [2.12 to 3.03] | 2.8 [2.36 to 3.31] | 2.6 [2.19 to 3.09]
Statistical Analysis 1: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous bisglycinate chelate 60 mg 1 twice-daily at Week 2; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.29 to 0.17]
Statistical Analysis 2: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous bisglycinate chelate 60 mg 1 twice-daily at Week 4; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.1, 95% CI [-0.57 to 0.31]
Statistical Analysis 3: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous bisglycinate chelate 60 mg 1 twice-daily at Week 6; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.75 to 0.46]
Statistical Analysis 4: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous bisglycinate chelate 60 mg 1 twice-daily at Week 8; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.05 to 0.53]
Statistical Analysis 5: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous ascorbate 100mg 1 once-daily at Week 2; Test type: Superiority or Other; p = 0.490, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.35 to 0.09]
Statistical Analysis 6: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous ascorbate 100 mg 1 once-daily at Week 4; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.58 to 0.29]
Statistical Analysis 7: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous ascorbate 100 mg 1 once-daily at Week 6; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.68 to 0.51]
Statistical Analysis 8: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Once-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 once-daily vs. Ferrous ascorbate 100 mg 1 once-daily at Week 8; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.84 to 0.72]
Statistical Analysis 9: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 twice-daily vs. Ferrous ascorbate 100mg 1 once-daily at Week 2; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.29 to 0.15]
Statistical Analysis 10: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 twice-daily vs. Ferrous ascorbate 100 mg 1 once-daily at Week 4; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.45 to 0.42]
Statistical Analysis 11: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 twice-daily vs. Ferrous ascorbate 100 mg 1 once-daily at Week 6; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.53 to 0.65]
Statistical Analysis 12: Comparison: Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily vs Ferrous Ascorbate 100 mg 1 Once-daily; Ferrous bisglycinate chelate 60 mg 1 twice-daily vs. Ferrous ascorbate 100 mg 1 once-daily at Week 8; Test type: Superiority or Other; p = 1, Repeated Measure ANOVA model; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.58 to 0.98]

5. Secondary Outcome: Difference in Percentage of Participants With Gastrointestinal Side Effects During 8 Weeks Treatment With Ferrous Bisglycinate Chelate and Ferrous Ascorbate
Description: The comparison in percentage of participants with gastrointestinal side effects during 8 week treatment period is reported. Gastrointestinal side effects during 8 weeks treatment included abdominal discomfort, gastritis, nausea, dyspepsia, change in bowel habit, constipation, faeces discolored, diarrhea and flatulence.
Time Frame: Up to Week 8
Population: Intent to treat (ITT) population which comprised of all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily | Ferrous Ascorbate 100 mg 1 Once-daily
Number analyzed (Participants) | 89 | 91 | 90
Percentage of participants | 6.7 | 9.9 | 11.1

ADVERSE EVENTS:
Time Frame: Serious adverse events and non-serious adverse events data was collected from Week 2 (Visit 2) to Week 8 (end of study drug or Visit 5)
Description: Serious adverse events and non-serious adverse events are reported for the Intent-to-Treat (ITT) population which comprised of all participants who were randomized and received at least one dose of the study medication
Arm/Group | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily | Ferrous Ascorbate 100 mg 1 Once-daily
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/91 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/91 | 0/90
Other Adverse Events (participants affected / at risk) | 8/89 | 12/91 | 12/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferrous Bisglycinate Chelate 60 mg 1 Once-daily (N=89) | Ferrous Bisglycinate Chelate 60 mg 1 Twice-daily (N=91) | Ferrous Ascorbate 100 mg 1 Once-daily (N=90)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Edema at the site of blood collection (General disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2 | 4
Gastritis (Gastrointestinal disorders) | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 1
Change in bowel habit (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Faeces discolored (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.